CLINICAL TRIAL: NCT05098418
Title: Trends of Acute Intoxication in Poison Control Centre, Ain Shams University Hospitals From 2015-2019
Brief Title: Trends of Acute Intoxication in Poison Control Centre
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: MTI University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dalia Kamal Zaafar Ali, Lecturer of clinical pharmacology, MTI University
Other Study IDs: ASU11032
Record Dates: First submitted 2021-10-05; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Poison Drug; Poison;Medicinal;Wrong Drug; Poisoning
Keywords: food poisoning; insecticides; detergents; heavy metals
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; Poisoning; Foodborne Diseases | interventions — Poisons

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 2015: total number of poisoned patients in 2015, including their demographic data
  Interventions: Drug: Poison
- 2016: total number of poisoned patients in 2016, including their demographic data
  Interventions: Drug: Poison
- 2017: total number of poisoned patients in 2017, including their demographic data
  Interventions: Drug: Poison
- 2018: total number of poisoned patients in 2018, including their demographic data
  Interventions: Drug: Poison
- 2019: total number of poisoned patients in 2019, including their demographic data
  Interventions: Drug: Poison

INTERVENTIONS:
Drug: Poison — standard of care and propre antidotes will be provided for each poisoned patients in addition to gastric lavage and activated charcoal administration when it is applicable
  Other Names: different poisonous materials

SUMMARY:
the study aim to investigate the trend of poisoning and its causative agents among different egyption people ages between 2015 and 2019

DETAILED DESCRIPTION:
This study aim to report different types of intoxication, the significant ages that intend to accidently ingest poisons or commit suicide, and the most commonly used chemicals in toxication, showing different rautes of administration between the years 2015 and 2019

ELIGIBILITY:
Inclusion Criteria:

- all medical records for patients admitted to PCC-ASUH emergency departmentwith the diagnosis of acute intoxication from 2015 t0 2019

Exclusion Criteria:

- any cases of acute intoxication before 2015 or after the end of 2019 cases of chronic intoxications were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all medical records for patients admitted to PCC-ASUH emergency departmentwith the diagnosis of acute intoxication from 2015 to 2019. patients include male and female patients in any age
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
investigating different interventions used for all cases of poisoned people form 2015 till 2019 | 5 years
  different interventions used for the treatment of different admitted cases of poisong or their death were taken from hospitals reports of patients admitted to the centre from 2015 till 2019

CONTACTS AND LOCATIONS:
Overall Officials: Maha Wahdan, Study Director — Lecturer of community and occupational medicine, faculty of medicine, Ain shams university
Locations (1):
- poison control centre Ain shams university hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No